CLINICAL TRIAL: NCT00869401
Title: Phase I/Randomized Phase II Trial of Either Dasatinib or Placebo Combined With Standard Chemo-Radiotherapy for Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: Dasatinib or Placebo, Radiation Therapy, and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCTG-N0877; NCI-2009-01179 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000637854 (Registry Identifier: PDQ (Physician Data Query)); U10CA025224 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Dasatinib; Temozolomide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Phase II) dasatinib + radiation + temozolomide (Experimental): Patients receive concomitant chemotherapy and radiation for cycle one for a total of 42 days, then patients receive adjuvant chemotherapy 28-42 days post cycle one treatment. Patients receive only dasatinib post cycle 8 until progressive disease, unacceptable adverse events or refusal.
  Interventions: Drug: dasatinib; Drug: temozolomide; Radiation: radiation therapy
- Group 2 (Phase II) placebo + radiation + temozolomide (Active Comparator): Patients receive concomitant chemotherapy and radiation for cycle one for a total of 42 days, then patients receive adjuvant chemotherapy 28-42 days post cycle one treatment. Patients receive only placebo post cycle 8 until progressive disease, unacceptable adverse events or refusal.
  Interventions: Drug: temozolomide; Other: placebo; Radiation: radiation therapy

INTERVENTIONS:
Drug: dasatinib — Given orally
  Arms: Group 1 (Phase II) dasatinib + radiation + temozolomide
Drug: temozolomide — Given orally
Other: placebo — Given orally
  Arms: Group 2 (Phase II) placebo + radiation + temozolomide
Radiation: radiation therapy — Radiation therapy is performed as 30 fractions of 200 cGy for a total of 6000 cGy.

SUMMARY:
Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It may also make tumor cells more sensitive to radiation therapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. This randomized phase I/II trial is studying the best dose of dasatinib and to see how well it works compared with a placebo when given together with radiation therapy and temozolomide in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
This trial includes a phase I dose-escalation study and a double-blind randomized phase II trial for patients with newly diagnosed glioblastoma multiforme (GBM). Phase I will be a cohort of 3 dose-escalation trial of dasatinib in combination with radiation and concomitant temozolomide. Patients receive concomitant chemotherapy and radiation therapy for cycle one. Patients receive adjuvant chemotherapy 28-42 days post cycle one treatment. Patients receive only dasatinib post cycle 8 treatment until progressive disease, unacceptable adverse events or refusal.

Phase II will be a randomized trial with two treatment arms. Patients will be randomized at the time of registration at a ratio of 1:2 respectively to either standard therapy arm (continuous daily placebo prior, during and after standard radiotherapy/temozolomide followed by temozolomide. For more information please see the Arms section. The primary objectives are listed below.

Primary Objectives:

1. To establish a maximum tolerated dose of dasatinib combined with radiation and temozolomide in this patient population (Phase I)
2. To determine the efficacy of dasatinib in combination with radiotherapy and concomitant and adjuvant temozolomide in patients with newly diagnosed glioblastoma, and compare it with the standard of care approach in the treatment of these patients consisting of radiotherapy and temozolomide, followed by adjuvant temozolomide (Phase II)

Patients are followed for 5 years post treatment. The study permanently closed to accrual on January 31, 2014.

ELIGIBILITY:
Pre-registration Inclusion Criteria:

1. Central Pathology Review - Central pathology review submission. This review is mandatory prior to registration to confirm eligibility.

Registration Inclusion Criteria:

1. Age ≥ 18 years
2. Histological Confirmation of Glioblastoma - Histologically confirmed newly diagnosed glioblastoma (GBM) (grade 4 astrocytoma) as determined by pre-registration central pathology review. Note: GBM with oligodendroglial features are not permitted in this study if they are 1p19q codeleted. Sites submitting GBM with oligodendroglial features will be asked to provide results of 1p/19q codeletion status.
3. Measurable or Evaluable Disease - Measurable or evaluable disease by gadolinium MRI or contrast CT scan. Note: Patients who have had a gross total resection are eligible on the basis of evaluable disease.
4. ECOG Performance Status 0, 1 or 2.
5. Required Laboratory Values:

   The following laboratory values obtained ≤ 14 days prior to registration.
   * Absolute neutrophil count (ANC) ≥ 1500/mm3
   * Platelet count ≥ 100,000/mm3
   * Hemoglobin > 9.0 g/dL
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * SGOT (AST) ≤ 2.5 x ULN
   * Creatinine ≤ 1.5 x ULN
6. Required INR Value: The following INR value obtained ≤ 28 days prior to registration

   * INR ≤ 1.5
7. Urine or Serum Pregnancy Test - Negative urine or serum pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only.
8. Written Informed Consent - Patient must provide written informed consent.
9. Return to Enrolling Institution - Patient must be willing to return to Alliance enrolling institution for follow-up.
10. Tissue Samples - Patient must be willing to provide tissue samples for research purposes.
11. Patient must be willing to provide tissue samples for research purposes.
12. Required Antibiotic Prophylaxis - Patient must be willing to comply with antibiotic prophylaxis with trimethoprim/sulfamethoxazole, pentamidine or dapsone.
13. Grapefruit and Grapefruit Juice - Patient must be willing to abstain from eating grapefruit or drinking grapefruit juice for the duration of the study treatment.
14. Ability to Swallow - Patient must have the ability to take oral medication (dasatinib must be swallowed whole).
15. Quality of Life (QOL) Questionnaires - Phase II patients only: Patients must be willing and able to complete QOL questionnaires independently or with the help of a caregiver.
16. Other Anti-Tumor Drug Therapies - Patient must be willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while being treated with dasatinib and temozolomide.

Registration Exclusion Criteria:

1. Pregnancy, Nursing and Required Contraception - Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential who are unwilling to employ adequate contraception throughout study treatment and for at least 12 weeks after study drug is stopped.
2. Prior Radiotherapy or Chemotherapy for Any CNS Neoplasm - Received any prior radiotherapy or chemotherapy for any CNS neoplasm (hormones, vitamins and growth factors are not considered chemotherapy for the purposes of this study.
3. Prior Surgery for Any CNS Neoplasm - Prior surgeries for any CNS neoplasms, other than surgery related to the current GBM diagnosis. Note: If Gliadel wafers are placed at time of primary resection, this would be considered prior therapy and patient would be ineligible.
4. Concurrent Illness or Disease - Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens. Including but not limited to:

   * History of bleeding diathesis
   * Current use of chronic systemic anticoagulation therapy that cannot be discontinued (antiplatelet agents, Aspirin)
   * Current chronic use of NSAIDs which cannot be discontinued
5. Pleural or Pericardial Effusions - Pleural or pericardial effusion of any grade.
6. Immunocompromised Status - Immunocompromised patients (other than that related to the use of corticosteroids) and patients known to be HIV positive and currently receiving antiretroviral therapy. Note: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
7. Uncontrolled Intercurrent Illness - Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Other Investigational Agents - Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
9. Other Active Malignancies - Other active malignancy ≤ 5 years prior to registration.

   Exceptions: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. Note: If there is a history of prior malignancy, they must not be receiving other specific treatment other than hormonal therapy for their cancer.
10. History of Cardiac or Metabolic Conditions:

    * Myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
    * Diagnosed congenital long QT syndrome
    * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
    * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
    * Patients with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration.
11. Clinically Significant Cardiovascular Disease - Patients may not have any clinically significant cardiovascular disease including the following:

    * Myocardial infarction or ventricular tachyarrhythmia within 6 months.
    * Ejection fraction less than institutional normal
    * Major conduction abnormality (unless a cardiac pacemaker is present)

    Note: Patients with any cardiopulmonary symptoms of unknown cause (e.g., shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to ECG to rule out QTc prolongation. The patient may be referred to a cardiologist at the discretion of the principal investigator.

    Patients with underlying cardiopulmonary dysfunction should be excluded from the study.
12. Congestive Heart Failure - New York Heart Association classification ≥ Class II Congestive Heart Failure.
13. Prohibited or Restricted Concomitant Treatments - Currently taking one of the following medications:

    * Enzyme inducing anti-convulsants (EIACs) Note: To be eligible, patient must be switched to non-EIAC medications ≥7 days prior to registration. See protocol for a list of EIAC and non-EIAC medications.
    * Potent inhibitors of CYP3A4 which cannot be discontinued. See protocol for a list of medications known to inhibit CYP3A4.
    * Medications known to prolong QT interval which cannot be discontinued or switched. See Appendix II for a list of medications which are known to prolong the QT interval.
    * Medications that may possibly prolong QT interval and produce a QTc that is ≥ 60 msec or a QTcF that is ≥ 450 msec. See Appendix II for a list of medications that may possibly prolong QTc.
    * St. John's Wort
    * H2 blockers or proton pump inhibitors (PPIs), such as famotidine (Pepcid) and omeprazole (Prilosec) respectively, which cannot be discontinued or switched to locally acting agents, such as Maalox, Mylanta and TUMS.
14. Allergy to Antibiotic Prophylaxis Medications - Severe allergy to sulfa medications and dapsone and pentamidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia N. Laack, MD, Study Chair — Mayo Clinic
Locations (207):
- United States (207):
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Greer Radiation Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin

REFERENCES:
- [Derived] Breen WG, Dixon JG, Anderson SK, Sarkaria JN, Brown PD, Yan ES, Kizilbash S, Galanis E, Anderson D, Tran D, Mazurczak M, Johnson DR, Geoffroy FJ, Leinweber C, Laack NN. Final report on North Central Cancer Treatment Group N0877 (alliance): A phase II randomized, placebo-controlled trial of chemoradiotherapy with or without dasatinib for glioblastoma. Neuro Oncol. 2025 Oct 1;27(10):2661-2670. doi: 10.1093/neuonc/noaf156. PMID 40579995

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 0 Phase I: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib at 50 mg twice a day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 100 mg/day until progression.
- Dose Level 0-A Phase I: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib at 100 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 100 mg/day until progression.
- Dose Level 1 Phase I: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib at 150 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 150 mg/day until progression.
- Group 1 (Phase II) Dasatinib + Radiation + Temozolomide: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib 150 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 150 mg/day until progression.
- Group 2 (Phase II) Placebo + Radiation + Temozolomide: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Placebo 150 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Placebo. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Placebo 150 mg/day until progression.
Period: Overall Study
Arm/Group | Dose Level 0 Phase I | Dose Level 0-A Phase I | Dose Level 1 Phase I | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide | Group 2 (Phase II) Placebo + Radiation + Temozolomide
Started | 3 | 3 | 7 | 138 | 66
Completed | 3 | 3 | 7 | 133 | 63
Not Completed | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Per protocol, the 8 canceled patients are excluded from all analysis
Groups:
- Phase I: All patients included in the Phase I portion of the study were published together for this results portion.
- Total: Total of all reporting groups
Arm/Group | Phase I | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide | Group 2 (Phase II) Placebo + Radiation + Temozolomide | Total
Number analyzed (Participants) | 13 | 133 | 63 | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (12.9) | 56.8 (11) | 58.2 (11.3) | 58 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 52 | 23 | 79
  Male | 9 | 81 | 40 | 130
Region of Enrollment [Number; unit: participants]
  United States | 13 | 133 | 63 | 209

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) is the primary endpoint and is defined as the time from study registration to time of death due to any cause. All patients who meet the eligibility criteria, have signed a consent form, and have received at least one dose of the regimens will be considered evaluable. Patients who are lost to follow-up will be censored at the date of their last follow-up. Patients still alive at the time of analysis will be censored. Only Phase II was evaluated for survival
Time Frame: Up to 5 years post treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide | Group 2 (Phase II) Placebo + Radiation + Temozolomide
Number analyzed (Participants) | 138 | 66
Months | 15.6 [14.4 to 19.6] | 19.3 [16.1 to 21.7]
Statistical Analysis 1: Comparison: Group 1 (Phase II) Dasatinib + Radiation + Temozolomide vs Group 2 (Phase II) Placebo + Radiation + Temozolomide; Test type: Superiority or Other; p = .222, Log Rank — Using Logrank Test; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.54 to 1.16]

2. Primary Outcome: The Number of Dose Limiting Toxicities(DLT) in Order to Determine Maximum Tolerable Dose(MTD) of Dasatinib Combined With Radiation and Temozolomide in This Patient Population.
Description: Doselimiting toxicity will be defined as: Adverse event at least possibly related to the study medication. All by CTCAE v3.0 criteria: Greater than or equal to grade 3: diarrhea or skin rash or desquamation or (other) clinically relevant non-hematological adverse event or non-hematologic adverse event at least possibly due to drug therapy. Or greater than or equal to grade 4: neutropenia or leukopenia or thrombocytopenia or radiation dermatitis or hematologic adverse event OR failure to administer greater than 75% of dasatinib TMZ or interruption of RT for more than 5 days due to adverse events.OR severe acute central nervous system deterioration attributable to TMZ, RT and or dasatinib which cannot be controlled with corticosteroid administration. The MTD for this study will be defined as the highest safely tolerated dose level where at most 1 out of 6 patients experience DLT with the next higher dose having at least 2 patients out of a maximum of 6 patients experience DLT.
Time Frame: Every cycle from first dose to end of rest period prior cycle 3
Population: Only Phase I patients were evaluated for maximum tolerable dose.
Measure: Number; unit: participants with Dose Limiting Toxicits
Arm/Group | Dose Level 0 Phase I | Dose Level 0-A Phase I | Dose Level 1 Phase I
Number analyzed (Participants) | 3 | 3 | 7
participants with Dose Limiting Toxicits | 1 | 0 | 1

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from study registration to the date of first observation of disease progression or death due to any cause (whichever comes first). If a patient has not progressed or died, progression-free survival is censored at the time of last follow-up. Only Phase II patients were evaluated for Progression-free survival
Time Frame: Up to 5 years post treatment
Population: All patients meeting the eligibility criteria that have signed a consent form and begun treatment will be considered evaluable
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide | Group 2 (Phase II) Placebo + Radiation + Temozolomide
Number analyzed (Participants) | 138 | 66
Months | 6.2 [4.4 to 8.2] | 7.8 [6.5 to 10.9]
Statistical Analysis 1: Comparison: Group 1 (Phase II) Dasatinib + Radiation + Temozolomide vs Group 2 (Phase II) Placebo + Radiation + Temozolomide; Test type: Superiority or Other; p = 0.183, Log Rank; Hazard Ratio (HR) = 0.806, 95% CI 2-sided [0.59 to 1.11]

4. Secondary Outcome: Objective Response
Description: Objective response to treatment will be determined by a combination of the results of neurological exam and the MRI and/or CT measurement of the tumor at each evaluation as is used for all NCCTG neuro-oncology trials. The proportion of patients in each response category will be summarized. Only phase II patients were evaluated for response.
Time Frame: Up to 5 years post treatment
Population: Participants that have at least one disease evaluation for assessing best response to treatment.
Measure: Number; unit: Proportion of participants
Arm/Group | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide | Group 2 (Phase II) Placebo + Radiation + Temozolomide
Number analyzed (Participants) | 98 | 48
Proportion of participants
  Progression | .31 | .19
  Stable | .59 | .73
  REGR | .08 | .02
  Partial Response | .02 | .06
  Complete Response | 0 | 0

ADVERSE EVENTS:
Groups:
- Dose Level 0 Phase I: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib at 100 mg twice a day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 100 mg/day until progression.
- Dose Level 0-A Phase I: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib at 100 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib100 mg/day until progression.
- Dose Level 1 Phase1: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib at 150 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 150 mg/day until progression.
- Group 2 (Phase II) Placebo + Radiation + Temozolomide: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Dasatinib 150 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Dasatinib. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Dasatinib 150 mg/day until progression.
- Group 1 (Phase II) Dasatinib + Radiation + Temozolomide: Cycle 1: Radiation therapy (RT) 60 Gy (2 Gy x 30 fractions) 5 days/week on weekdays for 6 weeks. Temozolomide (TMZ) 75 mg/m2/day and Placebo 150 mg/day starting with, and continuing through, RT. Cycle 2: 4-6 week rest period post RT/TMZ/Placebo. Cycles 3-8: (28-day cycles): TMZ 150 mg/m2 days 1-5 of cycle 3 and 200 mg/m2 days 1-5 of cycles 4-8. Cycle 3+: Placebo 150 mg/day until progression.
Arm/Group | Dose Level 0 Phase I | Dose Level 0-A Phase I | Dose Level 1 Phase1 | Group 2 (Phase II) Placebo + Radiation + Temozolomide | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 0/7 | 52/133 | 23/63
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 133/133 | 62/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 Phase I (N=3) | Dose Level 0-A Phase I (N=3) | Dose Level 1 Phase1 (N=7) | Group 2 (Phase II) Placebo + Radiation + Temozolomide (N=133) | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 5 (6)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 12 (13) | 8 (11)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 5 (6) | 8 (9)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 Phase I (N=3) | Dose Level 0-A Phase I (N=3) | Dose Level 1 Phase1 (N=7) | Group 2 (Phase II) Placebo + Radiation + Temozolomide (N=133) | Group 1 (Phase II) Dasatinib + Radiation + Temozolomide (N=63)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (12) | 2 (10) | 6 (37) | 107 (379) | 41 (135)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Hearing test abnormal (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 42 (61) | 13 (16)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (10) | 5 (13) | 91 (205) | 41 (107)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 7 (8)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (5) | 2 (2) | 3 (4) | 56 (97) | 25 (50)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
General symptom (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 27 (39) | 15 (22)
Leukocyte count decreased (Investigations) | 1 (2) | 2 (5) | 5 (13) | 67 (159) | 34 (149)
Lymphocyte count decreased (Investigations) | 2 (10) | 3 (14) | 7 (32) | 83 (217) | 46 (236)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (5) | 1 (4) | 47 (96) | 18 (53)
Platelet count decreased (Investigations) | 2 (7) | 2 (4) | 6 (19) | 80 (211) | 41 (131)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 4 (11)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 24 (25) | 9 (13)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 11 (15) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 4 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 4 (6)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Short stature (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 21 (33) | 8 (14)
Intracranial hemorrhage (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (15) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (4) | 44 (89) | 15 (28)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 33 (68) | 10 (23)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 2 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 3 (5) | 51 (96) | 19 (37)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (8)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes